CLINICAL TRIAL: NCT05148338
Title: The Effectivity of Lifestyle Interventions and Prevention in Patients With Atrial Fibrillation Referred for Ablation; a Randomized Controlled Trial
Brief Title: Prevention to Improve Outcomes After PVI
Acronym: POP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Lukas Dekker, Lukas Dekker, MD PhD, Principal Investigator, Clinical Professor, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZE2021.53
Record Dates: First submitted 2021-10-25; First posted 2021-12-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation; Risk Reduction; Nurse's Role
Keywords: pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation; Risk Reduction Behavior | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk intervention group (Experimental): Comprehensive risk factor management at specialized AF outpatient clinic concerning blood pressure, cholesterol, glycaemic control, physical inactivity, weight control, smoking, alcohol intake and sleep apnea.
  Interventions: Other: Comprehensive risk factor treatment
- Control group (Active Comparator): Standard of care. Treatment by cardiologist conform existing guidelines.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Comprehensive risk factor treatment — 1. Apnea screening with Home Sleep Apnea Test. Referral to sleep physician if apnea-hypopnea index (AHI) is greater than 5
  2. Weight management counseling by dietician if body mass index (BMI) is above 27 kg/m2
  3. Physical activity program under supervision of physiotherapist at a specialized cardiac rehabilitation centre if BMI is over 27 or if there are complaints during exercise
  4. Smoking cessation at specialized outpatient clinic
  5. Blood pressure control, lipid management, glycaemic control, alcohol intake reduction by specialized AF nurse
  6. Motivation and education through a digital health platform
  Arms: Risk intervention group
Other: Standard of care — Standard usual care: Treatment by cardiologist conform existing guidelines
  Arms: Control group

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia and has a rising prevalence due to an aging population. AF increases the patient's risk of hospitalization, heart failure and stroke and results into deterioration of quality of life. Treatment of symptomatic AF consists of either antiarrhythmic medication or a pulmonary vein isolation (PVI) catheter ablation. However, lots of patients experience recurrence of AF in the first year after PVI.

Previous studies showed that PVI outcomes depend on the presence of different treatable risk factors that influence the substrate for AF. Those risk factors include obesity, hypertension, cholesterol, diabetes mellitus, alcohol use, smoking and obstructive sleep apnea syndrome. However, research into the effect of treatment of those risk factors mainly consists of observational studies. Currently, it is not clear to what extent patients will benefit from comprehensive risk factor treatment prior to PVI in terms of ablation success and quality of life.

The aim of the current randomized controlled trial is to determine the effect of a nurse-led, technology-supported, personalized care pathway on hospital admissions for cardioversions and re-ablation in patients with AF that are referred for ablation.

Patients included in this study will be randomized to either the intervention group receiving the comprehensive risk treatment before PVI or the control group receiving standard usual care. Patients in the intervention group will visit the specialized AF nurse outpatient clinic and receive a personalized treatment plan (with a maximal duration of 6 months) including lifestyle interventions and medication. This includes sleep apnea screening with a Home Sleep Apnea Test (WatchPAT). Patients will also use the VitalHealth Engage platform. The digital platform can be used at home to report AF complaints, send home measurement and complete questionnaires. Furthermore, it supports the nurse in administering effective lifestyle changes by offering the patient personalized content and education.

Both study groups will be followed up to 12 months after ablation, during which hospital admissions for cardioversion and re-ablation are evaluated. At baseline, AFEQT, EQ5D and TBQ quality of life questionnaires will be performed. The questionnaires will be repeated prior to ablation, at 3 and 12 months after ablation. At baseline, pre-ablation and after 12 months laboratory tests (such as cholesterol) will be performed to evaluate adherence to lifestyle interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with paroxysmal or persistent symptomatic atrial fibrillation referred for initial catheter ablation
* Patients should be native Dutch speakers
* Patients are able to use the VitalHealth Engage platform on their own preferred device (tablet, mobile phone, computer)
* The patient has at least one of the following risks

  1. BMI ≥27 kg/m2,
  2. hyperlipidaemia (LDL-cholesterol >2.6 mmol/L or total cholesterol >5.0 mmol/L),
  3. hypertension (blood pressure >130/90 mmHg),
  4. diabetes mellitus with HbA1c ≥53 mmol/mol,
  5. active smoking,
  6. excess alcohol use (>14 equivalent units of alcohol / week)

Exclusion Criteria:

* Longstanding persistent atrial fibrillation (persistent AF for more than 1 year)
* Permanent atrial fibrillation
* Asymptomatic atrial fibrillation
* Prior catheter ablation
* Paroxysmal atrial fibrillation consisting of one episode with a reversible cause (e.g. fever, surgery, thyroid crisis, ischemic)
* Severe valvular heart disease
* Prior or soon foreseen implantation of cardiac device such as pacemaker or internal cardioverter defibrillator
* Unstable heart failure New York Heart Association (NYHA) IV, or heart failure necessitating admission <3 months before inclusion
* Cardiac surgery <3 months before inclusion or planned cardiac surgery
* Patient is not willing to use a mobile phone application or willing to undergo elaborate monitoring.
* Malignancy
* Life expectancy <1 year
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2025-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Number of hospital visits for cardioversion of AF and re-ablations | Up to 12 months after ablation or finishing risk treatment
  All events that occur between study inclusion and up to 12 months after ablation, including events prior to ablation. This means that events during the risk factor treatment period are also included

SECONDARY OUTCOMES:
Number of hospital visits for cardioversion of AF | Up to 12 months after ablation or finishing risk treatment
  All events that occur between study inclusion and up to 12 months after ablation, including events prior to ablation.
Number of reablations | Up to 12 months after ablation or finishing risk treatment
  All events that occur between study inclusion and up to 12 months after ablation, including events prior to ablation.
The composite of mortality, stroke or hospitalization for heart failure or acute ischemic events. | Up to 12 months after ablation
  Number of events. All events that occur between study inclusion and up to 12 months after ablation, including events prior to ablation.
All-cause mortality | Up to 12 months after ablation or finishing risk treatment
  Any deaths occurring during the study.
Number of strokes | Up to 12 months after ablation or finishing risk treatment
  All events that occur between study inclusion and up to 12 months after ablation, including events prior to ablation.
Hospitalizations for heart failure or acute ischemic events | Up to 12 months after ablation or finishing risk treatment
  Number of events. All events that occur between study inclusion and up to 12 months after ablation, including events prior to ablation.
Quality of Life - EQ-5D | Up to 12 months after ablation or finishing risk treatment
  Quality of Life as measured by the EuroQol 5 Dimensions (EQ-5D) questionnaire. The questionnaire compromises 5 dimensions describing different aspects of health and an overall health perception. The 5 dimensions can each be scored from level 1 to 5. Lower levels correspond with higher quality of life and higher levels correspond with lower quality of life. Overall health perception is scored with a visual analogue scale (VAS) ranging from 0 to 100, with lower values corresponding with worse outcomes and higher values corresponding to better outcomes.
Quality of Life - Atrial Fibrillation Effect on QualiTy of life survey (AFEQT) | Up to 12 months after ablation or finishing risk treatment
  Quality of Life as measured by the AFEQT questionnaire. The questionnaire contains 21 questions on a seven point Likert scale. Overall score ranges from 0 to 100. A score of 0 corresponds with complete disability, while a score of 100 corresponds with no disability.
Treatment burden - Treatment Burden Questionnaire (TBQ) | Up to 12 months after ablation or finishing risk treatment
  Treatment burden is the perception of cumulative work a patient has to perform to manage their health. The TBQ consists out of 15 items with a ten point rating scale. A higher score corresponds to a greater burden, while a lower score corresponds with a lower burden.
Rate of Success for ablation | From 3 months after ablation up to 12 months after ablation
  The ablation is considered to be successful if patients could stop their antiarrhythmics after 3 months (the blanking period) without recurrent arrhythmia. If patients develop recurrent arrhythmia and had to restart antiarrhythmics after the blanking period, the index ablation is considered unsuccessful.
Number of Cancellations of index ablation | Up to 12 months after finishing risk factor treatment
  Patients might experience absence of AF complaints after they have had effective treatment of their risk factors. The treating cardiologist might decide to cancel the index ablation if patients do not experience any AF complaints.

OTHER OUTCOMES:
Medical costs | Up to 12 months after ablation or finishing risk treatment
  An economic evaluation will be performed by examining all study intervention and AF related hospital costs. The total costs for both study groups will be compared
Cost-effectiveness ratio | Up to 12 months after ablation or finishing risk treatment
  Cost-effectiveness ratio will be analyzed by aggregating number of cardioversions and number of re-ablations and AF related medical costs. The cost-effectiveness ratio is the net costs per prevented cardioversion or re-ablation.
Patient value | Up to 12 months after ablation or finishing risk treatment
  Patient value will be assessed from a Value-Based Healthcare perspective. This will be done by dividing patient relevant outcomes, the quality of life as assessed by EQ-5D and AFEQT, through the costs per patient to achieve these outcomes.
Ablation - procedure times | During ablation
  Procedure time and fluoroscopy time
Ablation - DAP | During ablation
  Dose area product (DAP) during ablation, presented in mGy·cm2
Weight target achievement | Up to 12 months after finishing risk factor treatment
  Weight (in kg) will be measured at follow-up to determine whether patients did reach the target of losing 10% of total body weight.
Blood pressure target achievement | Up to 12 months after finishing risk factor treatment
  Blood pressure (in mmHg) will be measured at follow-up to determine whether the target of <130/80 mmHg was reached.
Success of treatment of sleep apnea | Up to 12 months after finishing risk factor treatment
  The apnea-hypopnea index (AHI) is used to determine the effect of sleep apnea treatment. AHI is determined at the start and end of sleep apnea treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Dekker, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermeer J, Vinck T, de Louw B, Slingerland S, van 't Veer M, Regis M, Jansen JM, van den Heuvel E, Dekker L. Improving outcomes of AF ablation by integrated personalized lifestyle interventions: rationale and design of the prevention to improve outcomes of PVI (POP) trial. Clin Res Cardiol. 2023 Jun;112(6):716-723. doi: 10.1007/s00392-023-02185-5. Epub 2023 Mar 31. PMID 37000245